CLINICAL TRIAL: NCT03941652
Title: Usability Study of the Sensors and the eMOM GDM Application eHealth in Treatment of Gestational Diabetes - eMOM GDM -Study
Brief Title: Usability Study of the Sensors and eMOM GDM Application
Acronym: eMOMGDM
Status: Active, not recruiting | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Business Finland (Other); Aalto University (Other); University of Helsinki (Other); Fujitsu Finland Oy (Unknown); Elisa Oyj (Unknown); CleverHealth Network (Unknown)
Responsible Party: Principal Investigator, Saila Koivusalo, Adjunct prof, Obstetrician, Development Manager, Helsinki University Central Hospital
Other Study IDs: HUS/2165/2018
Record Dates: First submitted 2019-04-25; First posted 2019-05-08 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Gestational Diabetes
Keywords: Gestational Diabetes; Continuous Glucose Values; Physical Activity; Nutrition; Behaviour Change; Stress; Recovery; Human-Computer Interaction (HCI); Mobile Application; Diet; Self-tracking; User interface; Health care professionals
MeSH Terms: conditions — Diabetes, Gestational; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (4):
- Women with gestational diabetes without a prior GDM: The investigators will evaluate the usability of the sensors and define what features the application should have and how the data should be presented to the users. Participants (n=up to 10) use the sensors for one week and fill out logbooks for physical activity, sleep and diet. Participants fill questionnaires before and after the usage period, and take part in semi-structured interview.
- Women with gestational diabetes with or without a prior GDM: The investigators define major usability issues with different versions of functional prototypes of eMOM GDM application developed in the project before moving to phase 2 of the study. GDM women (n=up to 12) will use the available version of the application for one week, and afterward the participants with GDM will take part in semi-structured interview.
- General pregnant women: The investigators will define major usability issues with different versions of functional prototypes of eMOM GDM application developed in the project before moving to phase 2 of the study. General pregnant women (n=up to 30) will use the available version of the application for one week, and afterward the general pregnant women will fill out a web form of usability of the application after the application week.
- Health care professionals: Nurses/midwifes (n=up to 20) will be interviewed for collecting user requirements for the professional eMOM GDM application in semi-structured interviews.

SUMMARY:
The principal aim of the eMOM GDM-project is to evaluate the effect of the eMOM GDM -application and the integrated service concept model on maternal and neonatal outcomes.

In the first phase of the project the investigators evaluate the usability, functionality and acceptability of developed eMOM GDM application and used sensors (continuous glucose meter, accelerometer, speech-enabled food record, optical pulse, beat-to-beat heart rate). Two different user interfaces (one for the women with GDM and one for the health care professionals) of the eMOM GDM application will we be developed and evaluated.

DETAILED DESCRIPTION:
The first phase of the eMOM GDM -project consists of two parts.

Phase 1.1. the usability of the sensors will be evaluated by asking participants with GDM diagnosis (n = up to 10) to use the sensors (Garmin Vivosmart 3, Medtronic Guardian Connect, Firstbeat Bodyguard 2, and Exced) and by collecting participants' blood glucose values from glucose meter (Contour Next ONE) for one week. Participants fill out a logbook for physical activity and sleeping for seven days, and a logbook for diet for three days during the study period. For ensuring the quality of food record a researcher will phone interview the participant based on her diet recordings.

Before starting using the sensors, the participants will fill Background questionnaire and Technology acceptance questionnaire (UTAUT). After the usage period, the participants will fill the same Technology acceptance questionnaire (UTAUT) and take part in semi-structured interview. The interview has to parts. In the first part, participants will be interviewed about the acceptability of sensors. In the second part, researcher will show a non-functional prototype of eMoM GDM application to the participant and will ask predetermined questions. Interview will be recorded and data obtained from the interviews will be transcribed for analysis.

Phase 1.2. will define major usability issues with different versions of functional prototypes of eMOM GDM application developed in the project before moving to phase 2 of the study. General pregnant women (n = up to 30 in total) and GDM women (n=up to 10) will use the available version of the application for one week, and afterward the participants with GDM will take part in semi-structured interview. Interview will be recorded and data will be transcribed for analysis. General pregnant women will fill out a web form of usability of the application after application week. Based on the responses of the form, the participants may be contacted for further inquiries about the usability issues they have reported. For ensuring the quality of food record a researcher will phone interview all participants based on her diet recordings.

In Phase 1.3 user requirements for the professional eMOM GDM application will be collected. The first aim of this evaluation is to define what features the application should have. These user requirements are collected with a semi-structured interview. Before the interview, background of the 15-20 nurses/midwifes is asked with background questionnaire on profession. In the interviews, the questions are predetermined, but some flexibility is allowed. Interviews will be recorded and data obtained from the interviews will be transcribed for analysis.

ELIGIBILITY:
Inclusion Criteria:

* General pregnant women at gestational week >=24
* GDM women without a prior GDM at gestational week >=24
* GDM women with or without a prior GDM at gestational week >=24

Exclusion Criteria:

* Type 1 Diabetes Mellitus
* Type 2 Diabetes Mellitus
* Use of medication that influences glucose metabolism in the beginning of the study (e.g. oral corticosteroids, metformin,insulin)
* Multiple Pregnancy
* Current substance abuse
* Severe psychiatric disorder
* Significant difficulty in cooperating (e.g. inadequate Finnish language skills)
* Significant physical disabilities

For health care professionals

Inclusion Criteria:

- Consult and treat women with GDM regularly

Exclusion Criteria:

- Inadequate Finnish language skills

Ages: 18 Years to 68 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — GDM can be studied only in pregnant women.
Study Population: * General population of pregnant women
  * Pregnant women without gestational diabetes in previous pregnancy
  * Pregnant women with or without gestational diabetes in previous pregnancies
  * Health care professionals (nurses/midwives)
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2019-05-27 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Basic version of the eMOM GDM application has developed | 1 week
  Goal of the eMOM GDM -project is develop an application for gestational diabetes. The basic version of eMOM GDM application is ready to use in Phase 2 when in all sectors of Software Usability Measurement Inventory (SUMI) scale have mean of 50 or higher during the same development period (sprint). SUMI is a rigorously tested and proven method of measuring software quality from the end user's point of view. Sectors which SUMI measures are efficiency, affect, helpfulness, control, learnability, and global usability of software.

SECONDARY OUTCOMES:
Acceptability of sensors assessed by UTAUT questionnaire | 1 week
  The acceptability of the sensors (Medtronic Guardian Connect, Garmin Vivosmart 3, Firsbeat Bodyguard 2, UKK Exsed, Ascensia Contour Next One) will be assessed by UTAUT (Unified Theory of Acceptance and Use of Technology)-questionnaire. UTAUT-questionnaire will be common for each sensor, so UTAUT will not be conducted for each sensor separately. The answers applied quantitative way so investigators are able analyzed change of acceptability of sensors caused by the intervention. Results applied to development of the eMOM GDM application.
Acceptability of sensors and eMOM GDM prototype application assessed by UTAUT questionnaire | 1 week
  The acceptability of the sensors (Garmin Vivosmart 3, Medtronic Guardian Connect, Ascensia Contour Next One, Speechgrinder Snackchat) and the eMOM GDM prototype application will be assessed by UTAUT (Unified Theory of Acceptance and Use of Technology) questionnaire. UTAUT questionnaire will be common for each sensor and the application, so UTAUT will not be conducted for each sensor separately. The answers applied quantitative way so investigators are able analyzed change of acceptability of sensors and application caused by the intervention. Results applied to development of the eMOM GDM application.
Usability of sensors and their current applications | 1 week
  Semi-structured interview of usability of chosen sensors and their current applications (Medtronic Guardian Connect, Garmin Vivosmart 3, Firsbeat Bodyguard 2, UKK Exsed, Ascensia Contour Next One).
  General questions related to the usability issues of sensors and their current applications.
  Sensors specific questions relate to usage of specific sensor and features of its application.
  The answers of participants give for investigators the guideline for development of eMOM GDM application. The answers itself won't be scaled, there isn't wrong or correct answers. Answers which repeat the most commonly in the interviews are the most common issues and they will have a higher priority in the guideline than answers which arises only in one interview.
First impressions of a partially functional prototype of the eMOM GDM | 1 week
  First impressions of eMOM GDM application questions relate to usability and acceptability of the eMOM GDM application which is under the development.
  The answers of participants give for investigators the guideline for development of eMOM GDM application. The answers itself won't be scaled, there isn't wrong or correct answers. Answers which repeat the most commonly in the interviews are the most common issues and they will have a higher priority in the guideline than answers which arises only in one interview.
Usability of eMOM GDM prototype application | 1 week
  Usability of the eMOM GDM prototype application will be assessed with a semi-structured interview. The interview has general questions about the usability issues of sensors (Garmin Vivosmart 3, Medtronic Guardian Connect, Ascensia Contour Next One, Speechgrinder Snackchat) and the eMOM GDM prototype application, and tasks which the participants try to solve using the eMOM GDM prototype application. The answers used as the guideline for development of eMOM GDM application.
Technical functionality of eMOM GDM application | 1 week
  Technical functionality of eMOM GDM application will be assessed by a web-based survey. The web-survey asks feedback from the eMOM GDM prototype application, and Garmin Vivosmart 3 bracelet, and there are 20 questions from Software Usability Measurement Inventory (SUMI) which the participant answers agree, disagree or not sure. This survey used as a guideline for development of eMOM GDM application. The answers tell how much major problems investigators still have in the eMOM GDM prototype application.
User requirements for professional eMOM GDM application | 2 hours
  User requirements will be collected through a semi-structured interviews. The interviews will be transcribed and a a framework analysis will be conducted to find the most important features. The answers used as the guideline for development of professional eMOM GDM application.

OTHER OUTCOMES:
Continuous glucose levels dataset | 1 week
  Dataset from Medtronic Guardian Connect glucose meter
Physical activity dataset | 1 week
  Dataset from Vivosmart 3, ExSed, Firstbeat Bodyguard 2, and physical activity logbook
Sleep dataset | 1 week
  Dataset from Vivosmart 3, Firstbeat Bodyguard 2, and sleep logbook
Recovery dataset | 1 week
  Dataset from Vivosmart 3 and Firstbeat Bodyguard 2
Stress dataset | 1 week
  Dataset from Vivosmart 3 and Firstbeat Bodyguard 2
Heart beat dataset | 1 week
  Dataset from Vivosmart 3 and Firstbeat Bodyguard 2
Nutrition dataset | 1 week
  Dataset from nutrition logbook

CONTACTS AND LOCATIONS:
Overall Officials: Seppo T Heinonen, prof, Study Director — Helsinki University Hospital, Women's Hospital
Locations (1):
- HUS, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kyto M, Koivusalo S, Tuomonen H, Stromberg L, Ruonala A, Marttinen P, Heinonen S, Jacucci G. Supporting the Management of Gestational Diabetes Mellitus With Comprehensive Self-Tracking: Mixed Methods Study of Wearable Sensors. JMIR Diabetes. 2023 Oct 31;8:e43979. doi: 10.2196/43979. PMID 37906216
- [Derived] Kyto M, Koivusalo S, Ruonala A, Stromberg L, Tuomonen H, Heinonen S, Jacucci G. Behavior Change App for Self-management of Gestational Diabetes: Design and Evaluation of Desirable Features. JMIR Hum Factors. 2022 Oct 12;9(4):e36987. doi: 10.2196/36987. PMID 36222806